CLINICAL TRIAL: NCT05633511
Title: Volumetric Changes of Soft Tissue Grafting. Comparison of Autologous PRF (Platelet-rich Fibrin ) & Autogenous CTG (Connective Tissue Grafts) . A Split-mouth Randomized Design
Brief Title: Changes of Soft Tissue Grafting: A Randomized Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003133
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): Participants will receive the CTG procedure on one side and the PRF procedure on the other. Both are standard of care soft tissue grafting methods and a split mouth design is standard of care.
  Interventions: Procedure: Split Mouth Design

INTERVENTIONS:
Procedure: Split Mouth Design — PRF on one side of mouth and CTG on the other side of participant's mouth.

SUMMARY:
To correct gum recession, patient's own tissue from the roof of the mouth is harvested and placed where there is root exposed. This is considered gold standard of treatment. Sometimes patient don't want to have second surgical site in their mouth and at the same time do not want to use alternative tissue from human or animal donor. Using patients' blood and preparing it as a membrane is the next best thing to correct gum recession.

DETAILED DESCRIPTION:
Patients that are interested in having corrective surgery for recession due to esthetic concerns or sensitivity will be enrolled in the study. The treatment site will randomly receive the procedure assignment. Intraoral scanner will be utilized to establish pre-op volume and will be repeated at each follow up visit. Total of 12 visits and 5 year duration is anticipated for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18yrs or older
2. Need of MG-tx for 2 or more sites for root coverage RT I and II (Cairo classification)
3. Class A +/-
4. No class V restoration present

Exclusion Criteria:

1. Patients who do not consent to recommended therapy
2. Patients who smoke
3. Patients who will not be able to comply with follow up protocols
4. Those who self report that they are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2035-12-30 (Estimated); Study Completion 2036-12-30 (Estimated)

PRIMARY OUTCOMES:
Compare autologous PRF & Autogenous CTG | 5 years
  Primary objective of this study is to compare in a split-mouth study the effectiveness of CTG vs. PRF in soft tissue augmentation and volume stability of each treatment modality in correcting the Cairo Class I, II defects in Periodontally affected patients

CONTACTS AND LOCATIONS:
Overall Officials: Tannaz Shapurian, DMD, MSc, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Nunn ME, Miyamoto T. Coronally advanced flaps (CAF) plus connective tissue graft (CTG) is the gold standard for treatment of Miller class I and II gingival defects. J Evid Based Dent Pract. 2013 Dec;13(4):157-9. doi: 10.1016/j.jebdp.2013.10.012. Epub 2013 Oct 11. No abstract available. PMID 24237738
- [Background] Padma R, Shilpa A, Kumar PA, Nagasri M, Kumar C, Sreedhar A. A split mouth randomized controlled study to evaluate the adjunctive effect of platelet-rich fibrin to coronally advanced flap in Miller's class-I and II recession defects. J Indian Soc Periodontol. 2013 Sep;17(5):631-6. doi: 10.4103/0972-124X.119281. PMID 24174758
- [Background] Chambrone L, Chambrone D, Pustiglioni FE, Chambrone LA, Lima LA. Can subepithelial connective tissue grafts be considered the gold standard procedure in the treatment of Miller Class I and II recession-type defects? J Dent. 2008 Sep;36(9):659-71. doi: 10.1016/j.jdent.2008.05.007. Epub 2008 Jun 26. PMID 18584934
- [Background] Natto ZS, Parashis AO, Jeong YN. Soft-Tissue Changes After Using Collagen Matrix Seal or Collagen Sponge With Allograft in Ridge Preservation: A Randomized Controlled Volumetric Study. J Oral Implantol. 2020 Dec 1;46(6):588-593. doi: 10.1563/aaid-joi-D-19-00080. PMID 32369569
- [Background] Tonetti MS, Cortellini P, Pellegrini G, Nieri M, Bonaccini D, Allegri M, Bouchard P, Cairo F, Conforti G, Fourmousis I, Graziani F, Guerrero A, Halben J, Malet J, Rasperini G, Topoll H, Wachtel H, Wallkamm B, Zabalegui I, Zuhr O. Xenogenic collagen matrix or autologous connective tissue graft as adjunct to coronally advanced flaps for coverage of multiple adjacent gingival recession: Randomized trial assessing non-inferiority in root coverage and superiority in oral health-related quality of life. J Clin Periodontol. 2018 Jan;45(1):78-88. doi: 10.1111/jcpe.12834. Epub 2017 Nov 21. PMID 29087001
- [Background] McLeod DE, Reyes E, Branch-Mays G. Treatment of multiple areas of gingival recession using a simple harvesting technique for autogenous connective tissue graft. J Periodontol. 2009 Oct;80(10):1680-7. doi: 10.1902/jop.2009.090187. PMID 19792859
- [Background] Keceli HG, Sengun D, Berberoglu A, Karabulut E. Use of platelet gel with connective tissue grafts for root coverage: a randomized-controlled trial. J Clin Periodontol. 2008 Mar;35(3):255-62. doi: 10.1111/j.1600-051X.2007.01181.x. Epub 2008 Jan 5. PMID 18190557
- See also: Evaluation of the effect of dose-dependent platelet-rich fibrin membrane on treatment of gingival recession: a randomized, controlled clinical trial — https://www.scielo.br/j/jaos/a/p54RtZLrf8gL4fTzSndJ57z/?lang=en